CLINICAL TRIAL: NCT05643885
Title: Cost Comparison Between Apixaban and Low Molecular Weight Heparin (LMWH) Among Venous Thromboembolism (VTE) Cancer Patients
Brief Title: A Study to Compare Health Care Costs Between Apixaban and Low Molecular Weight Heparin in Patients With Venous Thromboembolism and Cancer
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661183; NCT05643885 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- apixaban: patients treated with apixaban
- Low molecular weight heparin (LMWH): patients treated with low molecular weight heparin

SUMMARY:
The purpose of this study is to evaluate the health care resource utilization and costs associated with treating patients diagnosed with cancer and venous thromboembolism with apixaban or low molecular weight heparin. This is a retrospective database analysis of health care claims data. All-cause costs as well as costs associated with recurrent VTE, major bleeding, and clinically relevant nonmajor bleeding will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Venous thromboembolism (VTE) diagnosis between January 1 2017 and October 31 2021
* Evidence of active cancer
* At least 1 claim for apixaban or low molecular weight heparin (LMWH)
* Age 18 years or older

Exclusion Criteria:

* diagnosis of atrial fibrillation/flutter
* procedure for mechanical heart valve or inferior vena cava filter
* VTE diagnosis in the baseline period
* anticoagulant therapy in the baseline period
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active cancer who are newly diagnosed with venous thromboembolism (VTE) and treated with apixaban or low molecular weight heparin within 30 days following the VTE.
  Patients will be identified from the PharMetrics Plus health care claims database between the period of January 2017 and October 2021 if they have a VTE diagnosis and claim for apixaban or low molecular weight heparin during this time.
Sampling Method: Non-Probability Sample
Enrollment: 7304 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed venous thromboembolism (VTE) with active cancer who initiated apixaban or low molecular weight heparin (LMWH) within 30 days following VTE diagnosis were included in this study and data for eligible participants was retrospectively analyzed using IQVIA's database PharMetrics Plus.
Pre-assignment Details: The date of the first apixaban or LMWH prescription was considered as the index date. The analysis was conducted using retrospective data from 01 January 2016 through 31 December 2021. Available data was extracted and evaluated during 24 months of this retrospective observational study.
Groups:
- Apixaban: Participants with newly diagnosed VTE with active cancer who received apixaban within 30 days following the VTE diagnosis and no other anticoagulant (LMWH, other oral anti-coagulant [OAC], heparin or fondaparinux) between index VTE encounter date (first date of claim with a VTE diagnosis code) and the index date.
- LMWH: Participants with newly diagnosed VTE with active cancer who received LMWH within 30 days following the VTE diagnosis with a duration of at least 14 days and no apixaban or other anticoagulants between index VTE encounter and index date + 14 days.
Period: Overall Study
Arm/Group | Apixaban | LMWH
Started | 4299 | 3005
Completed | 4299 | 3005
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Apixaban: Participants with newly diagnosed VTE with active cancer who received apixaban within 30 days following the VTE diagnosis and no other anticoagulant (LMWH, other OAC, heparin or fondaparinux) between index VTE encounter date (first date of claim with a VTE diagnosis code) and the index date.
- Total: Total of all reporting groups
Arm/Group | Apixaban | LMWH | Total
Number analyzed (Participants) | 4299 | 3005 | 7304
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 29 | 54 | 83
  25-34 years | 75 | 79 | 154
  35-44 years | 234 | 239 | 473
  45-54 years | 802 | 621 | 1423
  55-64 years | 1951 | 1406 | 3357
  65-74 years | 799 | 458 | 1257
  >= 75 years | 409 | 148 | 557
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2119 | 1558 | 3677
  Male | 2180 | 1447 | 3627
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean All-Cause Healthcare Costs Per Participant Per Month (PPPM) for VTE Events
Description: The all-cause healthcare cost for VTE event was defined as the sum of total cost associated with the total inpatient, total outpatient, and total pharmacy costs for the VTE event. Costs were converted to 2021 United States dollars (USD) using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: From index date until health plan disenrollment, index therapy discontinuation, switch to another anticoagulant or end of study period (up to 72 months); data observed retrospectively over 24 months
Population: Analysis population included all participants whose data were included and observed in the study. Here, "Overall Number of Participants Analyzed" reflects the pseudo-population created using stabilized inverse probability of treatment weighting (IPTW). Hence, numbers are different here from those presented in participant flow and baseline section.
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 4288 | 3022
USD per participant per month | 16420 (23354) | 21312 (27337)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p < 0.0001, Weighted t-test

2. Primary Outcome: Mean All-Cause Healthcare Outpatient Pharmacy Costs PPPM for VTE Events
Description: The all-cause healthcare outpatient pharmacy cost for VTE event was defined as the total cost associated with the outpatient pharmacy costs for the VTE event. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: Analysis population included all participants whose data were included and observed in the study. Here, "Overall Number of Participants Analyzed" reflects the pseudo-population created using stabilized IPTW. Hence, numbers are different here from those presented in participant flow and baseline section.
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 4288 | 3022
USD per participant per month | 2452 (5376) | 2654 (4701)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p < 0.0001, Weighted t-test

3. Primary Outcome: Mean All-Cause Healthcare Outpatient Medical Costs PPPM for VTE Events
Description: The all-cause healthcare outpatient medical cost for VTE event was defined as the total cost associated with the outpatient medical costs (excluding pharmacy costs) for the VTE event. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 4288 | 3022
USD per participant per month | 8028 (11644) | 10042 (12759)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p < 0.0001, Weighted t-test

4. Primary Outcome: Mean All-Cause Healthcare Hospitalization Costs PPPM for VTE Events
Description: The all-cause healthcare hospitalization cost for VTE event was defined as the cost associated with the inpatient hospitalization for the VTE event. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 4288 | 3022
USD per participant per month | 5940 (17512) | 8616 (22667)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p < 0.0001, Weighted t-test

5. Primary Outcome: Mean All-Cause Healthcare Costs PPPM for Recurrent VTE Events
Description: Recurrent VTE was identified based on inpatient claims with VTE as the primary diagnosis on any claim (international classification of diseases, tenth revision, clinical modification [ICD-10-CM] diagnosis codes). Recurrent VTE all cause healthcare costs were defined as the costs associated with the first recurrent VTE hospitalization and all subsequent VTE costs in the inpatient (primary or secondary diagnosis) or outpatient (any position) setting. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: Analysis population included all participants whose data were included and observed in the study. Here, "Overall Number of Participants Analyzed" reflects the pseudo-population created using stabilized IPTW and who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 371 | 391
USD per participant per month | 11277 (19873) | 13074 (21342)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.2303, Weighted t-test

6. Primary Outcome: Mean All-Cause Healthcare Outpatient Medical Costs PPPM for Recurrent VTE Events
Description: Recurrent VTE was identified based on inpatient claims with VTE as the primary diagnosis on any claim (ICD-10-CM diagnosis codes). Recurrent VTE outpatient medical costs included costs associated with physician office visits, emergency room visits, laboratory or pathology visits, radiology exams, and outpatient surgical visits. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 371 | 391
USD per participant per month | 827 (2367) | 884 (2430)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.7403, Weighted t-test

7. Primary Outcome: Mean All-Cause Healthcare Hospitalization Costs PPPM for Recurrent VTE Events
Description: Recurrent VTE was identified based on inpatient claims with VTE as the primary diagnosis on any claim (ICD-10-CM diagnosis codes). The all-cause healthcare hospitalization cost for recurrent VTE event was defined as the cost associated with the inpatient hospitalization for the recurrent VTE event. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 371 | 391
USD per participant per month | 10450 (19670) | 12190 (21175)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.2414, Weighted t-test

8. Primary Outcome: Mean All-Cause Healthcare Costs PPPM for Major Bleeding Related VTE Events
Description: Major bleeding was defined by primary discharge diagnosis on any claim in the inpatient setting, including gastrointestinal (GI) bleeding, intracranial hemorrhage (ICH), and other major bleeding. Major bleeding-related all cause healthcare costs were defined as costs associated with the first major bleeding hospitalization plus all subsequent bleeding costs occurring in the inpatient (primary or secondary diagnosis) or outpatient setting (any position). Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 205 | 225
USD per participant per month | 19384 (30260) | 22719 (30865)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.2592, Weighted t-test

9. Primary Outcome: Mean All-Cause Outpatient Medical Costs PPPM for Major Bleeding Related VTE Events
Description: Major bleeding was defined by primary discharge diagnosis on any claim in the inpatient setting, including GI bleeding, ICH and other major bleeding. Major bleeding-related all cause outpatient medical costs were major bleeding related outpatient costs associated with physician office visits, emergency room visits, laboratory or pathology visits, radiology exams, and outpatient surgical visits. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 205 | 225
USD per participant per month | 268 (1021) | 346 (1256)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.4837, Weighted t-test

10. Primary Outcome: Mean All-Cause Hospitalization Costs PPPM for Major Bleeding Related VTE Events
Description: Major bleeding was defined by primary discharge diagnosis on any claim in the inpatient setting, including GI bleeding, ICH, and other major bleeding. Major bleeding-related all cause healthcare costs were defined as costs associated with the first major bleeding hospitalization plus all subsequent bleeding costs occurring in the inpatient (primary or secondary diagnosis). Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 205 | 225
USD per participant per month | 19116 (30241) | 22373 (30822)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.1355, Weighted t-test

11. Primary Outcome: Mean All-Cause Healthcare Costs PPPM for Clinically Relevant Non-Major (CRNM) Bleeding Related VTE Events
Description: CRNM bleeding-related all cause healthcare costs were combination of bleeding related inpatient and outpatient costs. CRNM bleeding was defined as an inpatient encounter with a secondary diagnosis code for bleeding (without a major bleeding code in the primary position) or an outpatient encounter with a diagnosis code in any position for CRNM GI bleeding or other non-critical types of bleeding. Any CRNM bleeding events that followed a major bleeding event were not included in the analysis of CRNM bleeding. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 907 | 777
USD per participant per month | 4883 (13142) | 5227 (14230)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.6066, Weighted t-test

12. Primary Outcome: Mean All-Cause Outpatient Medical Costs PPPM for CRNM Bleeding Related VTE Events
Description: CRNM bleeding was defined as an inpatient encounter with a secondary diagnosis code for bleeding (without a major bleeding code in the primary position) or an outpatient encounter with a diagnosis code in any position for CRNM GI bleeding or other non-critical types of bleeding. CRNM bleeding all cause outpatient medical costs were major bleeding related outpatient costs associated with physician office visits, emergency room (ER) visits, laboratory or pathology visits, radiology exams, and outpatient surgical visits. Any CRNM bleeding events that followed a major bleeding event were not included in the analysis of CRNM bleeding. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 907 | 777
USD per participant per month | 431 (1134) | 483 (1291)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.3795, Weighted t-test

13. Primary Outcome: Mean All-Cause Hospitalization Costs PPPM for CRNM Bleeding Related VTE Events
Description: CRNM bleeding was defined as an inpatient encounter with a secondary diagnosis code for bleeding (without a major bleeding code in the primary position) or an outpatient encounter with a diagnosis code in any position for CRNM GI bleeding or other non-critical types of bleeding. Any CRNM bleeding events that followed a major bleeding event were not included in the analysis of CRNM bleeding. Costs were converted to 2021 USD using the medical component of the consumer price index and was expressed as cost per participant per month. The date of the first apixaban or LMWH prescription on or within the 30 days following a VTE diagnosis was considered as the index date.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: USD per participant per month
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 907 | 777
USD per participant per month | 4452 (13126) | 4744 (14232)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.6618, Weighted t-test

14. Secondary Outcome: Mean Number of Hospitalizations Per Participant Per Month (PPPM) for VTE Events
Description: Mean number of hospitalizations PPPM for VTE events are reported in this outcome measure. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hospitalizations PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 1837 | 1663
Hospitalizations PPPM | 0.4 (0.4) | 0.4 (0.4)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.2337, Weighted t-test

15. Secondary Outcome: Mean Number of Outpatient Medical Visits PPPM for VTE Events
Description: Mean number of outpatient medical visits PPPM for VTE events are reported in this outcome measure. Outpatient visits included physician office visits, ER visits, laboratory or pathology visits, radiology exams, and outpatient surgical visits and ancillary or other services. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: Analysis population included all participants whose data were included and observed in the study. Here, "Overall Number of Participants Analyzed (N)" reflects the pseudo-population created using stabilized IPTW. Hence, numbers are different here from those presented in participant flow and baseline section. All participants reported under "N" contributed data to table; however, may not have evaluable data for every row. Number analyzed (n)= number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Outpatient medical visits PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 4288 | 3022
Outpatient medical visits PPPM
  Physician office visits: number analyzed (Participants) | 4183 | 2968
  Physician office visits | 3.0 (3.0) | 3.5 (3.1)
  ER only visits: number analyzed (Participants) | 1937 | 1640
  ER only visits | 0.2 (0.3) | 0.2 (0.4)
  laboratory or pathology visits: number analyzed (Participants) | 3987 | 2870
  laboratory or pathology visits | 5.6 (7.0) | 8.1 (9.5)
  Radiology: number analyzed (Participants) | 3647 | 2695
  Radiology | 1.6 (2.8) | 2.1 (3.1)
  Surgical services: number analyzed (Participants) | 2671 | 2104
  Surgical services | 0.4 (0.7) | 0.6 (0.8)
  Ancillary/other services: number analyzed (Participants) | 4151 | 2977
  Ancillary/other services | 6.5 (7.0) | 7.7 (7.1)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Physician office visits; Test type: Superiority; p < 0.0001, Weighted t-test
Statistical Analysis 2: Comparison: Apixaban vs LMWH; ER only visits; Test type: Superiority; p < 0.0001, Weighted t-test
Statistical Analysis 3: Comparison: Apixaban vs LMWH; laboratory or pathology visits; Test type: Superiority; p < 0.0001, Weighted t-test
Statistical Analysis 4: Comparison: Apixaban vs LMWH; Radiology; Test type: Superiority; p < 0.0001, Weighted t-test
Statistical Analysis 5: Comparison: Apixaban vs LMWH; Surgical services; Test type: Superiority; p < 0.0001, Weighted t-test
Statistical Analysis 6: Comparison: Apixaban vs LMWH; Ancillary/other services; Test type: Superiority; p < 0.0001, Weighted t-test

16. Secondary Outcome: Mean Number of Prescription Fills PPPM for VTE Events
Description: Mean number of prescription fills PPPM for VTE events are reported in this outcome measure. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Prescription fills PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 4287 | 3021
Prescription fills PPPM | 5.0 (4.1) | 5.6 (4.5)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p < 0.0001, Weighted t-test

17. Secondary Outcome: Mean Number of Hospitalizations PPPM for Recurrent VTE Events
Description: Recurrent VTE was identified based on inpatient claims with VTE as the primary diagnosis on any claim (ICD-10-CM diagnosis codes). Mean number of hospitalizations PPPM for recurrent VTE events are reported in this outcome measure. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hospitalizations PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 371 | 391
Hospitalizations PPPM | 0.6 (0.5) | 0.6 (0.5)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.7290, Weighted t-test

18. Secondary Outcome: Mean Number of Outpatient Medical Visits PPPM for Recurrent VTE Events
Description: Recurrent VTE was identified based on inpatient claims with VTE as the primary diagnosis on any claim (ICD-10-CM diagnosis codes). Outpatient visits included physician office visits, ER only visits, laboratory or pathology visits, radiology, and surgical services and ancillary or other services. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: Analysis population included all participants whose data were included and observed in the study. Here, "Overall Number of Participants Analyzed (N)" reflects the pseudo-population created using stabilized IPTW. All participants reported under "N" contributed data to table; however, may not have evaluable data for every row. Number analyzed (n)= number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Outpatient medical visits PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 371 | 391
Outpatient medical visits PPPM
  Physician office visits: number analyzed (Participants) | 186 | 204
  Physician office visits | 0.7 (1.7) | 0.6 (1.6)
  ER only visits: number analyzed (Participants) | 25 | 24
  ER only visits | 0.0 (0.1) | 0.0 (0.1)
  Laboratory or pathology visits: number analyzed (Participants) | 94 | 120
  Laboratory or pathology visits | 0.6 (1.8) | 0.8 (2.9)
  Radiology: number analyzed (Participants) | 71 | 83
  Radiology | 0.2 (0.6) | 0.2 (0.8)
  Surgical services: number analyzed (Participants) | 12 | 28
  Surgical services | 0.0 (0.1) | 0.0 (0.1)
  Ancillary or other services: number analyzed (Participants) | 143 | 167
  Ancillary or other services | 1.1 (3.5) | 0.7 (2.5)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Physician office visits; Test type: Superiority; p = 0.3686, Weighted t-test
Statistical Analysis 2: Comparison: Apixaban vs LMWH; ER only visits; Test type: Superiority; p = 0.2747, Weighted t-test
Statistical Analysis 3: Comparison: Apixaban vs LMWH; Laboratory or pathology visits; Test type: Superiority; p = 0.1049, Weighted t-test
Statistical Analysis 4: Comparison: Apixaban vs LMWH; Radiology; Test type: Superiority; p = 0.8425, Weighted t-test
Statistical Analysis 5: Comparison: Apixaban vs LMWH; Surgical services; Test type: Superiority; p = 0.9755, Weighted t-test
Statistical Analysis 6: Comparison: Apixaban vs LMWH; Ancillary or other services; Test type: Superiority; p = 0.0582, Weighted t-test

19. Secondary Outcome: Mean Number of Hospitalizations PPPM for Major Bleeding Related VTE Events
Description: Major bleeding was defined by primary discharge diagnosis on any claim in the inpatient setting, including GI bleeding, ICH and other major bleeding. Mean number of hospitalizations PPPM for recurrent VTE events are reported in this outcome measure. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hospitalizations PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 205 | 225
Hospitalizations PPPM | 0.6 (0.5) | 0.6 (0.5)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.9796, Weighted t-test

20. Secondary Outcome: Mean Number of Outpatient Medical Visits PPPM for Major Bleeding Related VTE Events
Description: Major bleeding was defined by primary discharge diagnosis on any claim in the inpatient setting, including GI bleeding, ICH and other major bleeding. Outpatient visits included physician office visits, ER only visits, laboratory or pathology visits, radiology, and surgical services and ancillary or other services. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Outpatient medical visits PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 205 | 225
Outpatient medical visits PPPM
  Physician office visits: number analyzed (Participants) | 59 | 86
  Physician office visits | 0.3 (0.9) | 0.5 (1.4)
  ER only visits: number analyzed (Participants) | 19 | 17
  ER only visits | 0.0 (0.1) | 0.0 (0.2)
  Laboratory or pathology visits: number analyzed (Participants) | 28 | 41
  Laboratory or pathology visits | 0.4 (1.6) | 0.3 (1.2)
  Radiology: number analyzed (Participants) | 25 | 16
  Radiology | 0.1 (0.3) | 0.0 (0.2)
  Surgical services: number analyzed (Participants) | 21 | 30
  Surgical services | 0.0 (0.2) | 0.1 (0.4)
  Ancillary or other services: number analyzed (Participants) | 28 | 43
  Ancillary or other services | 0.2 (0.9) | 0.3 (1.4)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Physician office visits; Test type: Superiority; p = 0.0379, Weighted t-test
Statistical Analysis 2: Comparison: Apixaban vs LMWH; ER only visits; Test type: Superiority; p = 0.9034, Weighted t-test
Statistical Analysis 3: Comparison: Apixaban vs LMWH; Laboratory or pathology visits; Test type: Superiority; p = 0.5452, Weighted t-test
Statistical Analysis 4: Comparison: Apixaban vs LMWH; Radiology; Test type: Superiority; p = 0.1644, Weighted t-test
Statistical Analysis 5: Comparison: Apixaban vs LMWH; Surgical services; Test type: Superiority; p = 0.0650, Weighted t-test
Statistical Analysis 6: Comparison: Apixaban vs LMWH; Ancillary or other services; Test type: Superiority; p = 0.3866, Weighted t-test

21. Secondary Outcome: Mean Number of Hospitalizations PPPM for CRNM Bleeding Related VTE Events
Description: CRNM bleeding was defined as an inpatient encounter with a secondary diagnosis code for bleeding (without a major bleeding code in the primary position) or an outpatient encounter with a diagnosis code in any position for CRNM GI bleeding or other non-critical types of bleeding. Mean number of hospitalizations PPPM for recurrent VTE events are reported in this outcome measure. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hospitalizations PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 907 | 777
Hospitalizations PPPM | 0.5 (0.4) | 0.5 (0.4)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Test type: Superiority; p = 0.5660, Weighted t-test

22. Secondary Outcome: Mean Number of Outpatient Medical Visits PPPM for CRNM Bleeding Related VTE Events
Description: CRNM bleeding was defined as an inpatient encounter with a secondary diagnosis code for bleeding (without a major bleeding code in the primary position) or an outpatient encounter with a diagnosis code in any position for CRNM GI bleeding or other non-critical types of bleeding. Outpatient visits included physician office visits, ER only visits, laboratory or pathology visits, radiology, and surgical services and ancillary or other services. Index date was defined as the date of the first apixaban or LMWH prescription claim on or within the 30 days following a VTE diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Outpatient medical visits PPPM
Arm/Group | Apixaban | LMWH
Number analyzed (Participants) | 907 | 777
Outpatient medical visits PPPM
  Physician office visits: number analyzed (Participants) | 479 | 426
  Physician office visits | 0.3 (0.7) | 0.4 (0.8)
  ER only visits: number analyzed (Participants) | 170 | 174
  ER only visits | 0.1 (0.2) | 0.1 (0.2)
  Laboratory or pathology visits: number analyzed (Participants) | 368 | 318
  Laboratory or pathology visits | 0.7 (1.9) | 0.9 (2.8)
  Radiology: number analyzed (Participants) | 185 | 158
  Radiology | 0.1 (0.5) | 0.1 (0.3)
  Surgical services: number analyzed (Participants) | 153 | 132
  Surgical services | 0.1 (0.2) | 0.1 (0.2)
  Ancillary or other services: number analyzed (Participants) | 273 | 271
  Ancillary or other services | 0.3 (1.0) | 0.4 (1.4)
Statistical Analysis 1: Comparison: Apixaban vs LMWH; Physician office visits; Test type: Superiority; p = 0.0425, Weighted t-test
Statistical Analysis 2: Comparison: Apixaban vs LMWH; ER only visits; Test type: Superiority; p = 0.8634, Weighted t-test
Statistical Analysis 3: Comparison: Apixaban vs LMWH; Laboratory or pathology visits; Test type: Superiority; p = 0.0399, Weighted t-test
Statistical Analysis 4: Comparison: Apixaban vs LMWH; Radiology; Test type: Superiority; p = 0.0996, Weighted t-test
Statistical Analysis 5: Comparison: Apixaban vs LMWH; Surgical services; Test type: Superiority; p = 0.7655, Weighted t-test
Statistical Analysis 6: Comparison: Apixaban vs LMWH; Ancillary or other services; Test type: Superiority; p = 0.1499, Weighted t-test

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be assessed or monitored during this study
Description: This observational retrospective study involved data that existed as structured data by the time of study start. In these data sources, individual participants data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participants, identifiable reporter, a suspect product, and event) was not met. Hence, adverse events were not assessed or evaluated which explains "0" participants at risk.
Arm/Group | Apixaban | LMWH
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT05643885/Prot_SAP_000.pdf